CLINICAL TRIAL: NCT05152940
Title: ERTU-SODIUM: Double-blind, Prospective, Randomized, Crossover, Placebo-control Study on the Effects of the SGLT2 Inhibitor Ertugliflozin on the Regulation of Interstitial Volume, Plasma Volume, Subcutaneous Sodium Storage, and the Functionality of the Subcutaneous Glycosaminoglycan Network in Patients With Heart Failure With Reduced Ejection Fraction (HFrEF)
Brief Title: ERTU-SODIUM: Study on the Effects of Ertugliflozin on Sodium Storage, Interstitial Volume, and Plasma Volume in HFrEF
Acronym: ERTU-SODIUM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Carlos Santos-Gallego, Principal Investigator, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PD21-12423
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Congestion
Keywords: SGLT2 inhibitors; heart failure with reduced ejection fraction; congestion; sodium
MeSH Terms: interventions — ertugliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ertugliflozin then Placebo (Active Comparator): Treatment with Ertugliflozin for one month, washout period for one month, and then with Placebo for one month
  Interventions: Drug: Ertugliflozin; Drug: Placebo
- Placebo (Active Comparator): Treatment with matching placebo for one month, washout period for one month, and then Ertugliflozin for one month
  Interventions: Drug: Ertugliflozin; Drug: Placebo

INTERVENTIONS:
Drug: Ertugliflozin — Treatment with Ertugliflozin 5 mg oral once per day for one month
Drug: Placebo — Treatment with matching placebo to ertugliflozin administered orally once daily for a period of one month

SUMMARY:
The overall hypothesis is that treatment with the SGLT2 inhibitor Ertugliflozin induces a differential regulation in interstitial fluid vs plasma volume, with more reduction of the volume from the interstitial fluid than from the circulating plasma volume, which results in Ertugliflozin inducing more potent congestion relief with minimal impact on blood volume and organ perfusion. Ertugliflozin reduces the levels of sodium and water from the skin and the interstitial tissue (which improves tissue congestion).

DETAILED DESCRIPTION:
The glucosaminoglycan (GAG) network in the subcutaneous interstitium can non-osmotically bind large amounts of sodium. Therefore, the GAG network creates a hypertonic sodium concentration without fluid accumulation. This means that the subcutaneous GAG act as a third compartment that is able to non-osmotically store sodium without inducing congestion, thus serving as buffer in the case of sodium overload.

The researchers hypothesize that the SGLT2 inhibitor Ertugliflozin enhances the functionality of the subcutaneous GAG network. The hypothesis is that Ertugliflozin-induced GAG functionality induces more potent congestion relief (reduction in sodium and water content in the interstitial tissue) with minimal impact on blood volume and organ perfusion.

The research team will perform a randomized clinical trial with a cross-over design. Patients with heart failure with reduced ejection fraction (HFrEF) will be randomized to the SGLT2 inhibitor Ertuglifozin or to placebo. Skin punch biopsy will be performed before treatment and after treatment (one month) to evaluate skin content of water and sodium. At each time point, an oral salt challenge will be performed to investigate the functionality of the GAG network, and whether Ertugliflozin mitigates the degree of tissue and vascular congestion after this oral salt challenge as compared with placebo.

The overall hypothesis is that treatment with the SGLT2 inhibitor Ertugliflozin induces a differential regulation in interstitial fluid vs plasma volume, with more reduction of the volume from the interstitial fluid than from the circulating plasma volume, which results in Ertugliflozin inducing more potent congestion relief with minimal impact on blood volume and organ perfusion. Ertugliflozin reduces the levels of sodium and water from the skin and the interstitial tissue (which improves tissue congestion). This overarching hypothesis causes:

1. in the baseline situation, chronic treatment with Ertugliflozin:

   1.1. will reduce skin/tissue congestion as demonstrated by lower skin water content and lower volume of interstitial-extracellular fluid

   1.2. will reduce skin sodium content due to a mobilization of sodium from the subcutaneous glucosaminoglycan (GAG) network

   1.3. will create a differential regulation of interstitial vs plasmatic volume, with ertugliflozin decreasing tissue congestion (B-lines and dielectric resistance in lungs) better than placebo

   1.4. will only cause a mild reduction in plasma volume with no neurohormonal activation

   1.5. will ameliorate GAG structure: higher GAG levels, higher sulfated (functional) GAG, less expression of enzymes degrading GAG, less GAG degradation products in plasma
2. after an oral salt challenge (sodium overload), previous chronic treatment with Ertugliflozin:

2.1. will improve the sodium buffering capacity of the skin GAG network, meaning ertugliflozin will enhance non-osmotic sodium storage in the skin without causing tissue congestion (edema) or vascular congestion (increase in plasma volume and filling pressures).

2.2. will reduce skin/tissue congestion (as mentioned in 2.1): lower skin water content and interstitial-extracellular fluid volume

2.3. will not cause vascular congestion, will not raise plasma volume or LV filling pressures

In summary, Ertugliflozin will protect HFrEF patients from acute decompensations induced by dietary transgressions by enhancing the skin sodium buffering capacity

ELIGIBILITY:
Inclusion criteria:

* age >18 years;
* males and females (females of child bearing potential must be using adequate contraceptive precautions)
* diagnosis of heart failure (New York Heart Association [NYHA] functional class II to III);
* Left ventricular ejection fraction <40%;
* stable symptoms and medical therapy within the last month.
* Informed consent has to be given in written form

Exclusion criteria:

* taking SGLT2i in the last month
* acute coronary syndrome or cardiac surgery within the last month;
* estimated glomerular filtration rate <20 ml/kg/min;
* use of continuous parental inotropic agents;
* systolic blood pressure <90 mm Hg;
* LVAD implantation or cardiac transplantation
* pregnant or lactating women; and
* any other medical condition considered unappropriated by a study physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in the skin water content | Baseline and One month
  Skin water content is measured as total (wet) weight - dry weight, determined after desiccation at 90°C for 24 hours to stable weight

SECONDARY OUTCOMES:
Change in skin sodium content | Baseline and One month
  Skin sodium content will be measured by flame spectrophotometry after dry ashing
Change in interstitial Fluid | Baseline and One month
  Interstitial Fluid to measure tissue congestion and will be calculated as Extracellular Volume minus Plasma Volume
Change in pulmonary fluid | Baseline and One month
  Pulmonary fluid content to measure tissue congestion and is quantified using remote dielectric sensing with ReDS Vest
Change in the number of pulmonary Kerley's B-lines | Baseline and One month
  The number of pulmonary Kerley's B-lines (aka "comets") to measure tissue congestion and will be quantified using lung ultrasound
Change in the plasma volume | Baseline and One month
  Plasma volume to measure vascular congestion.
Change in vascular congestion | Baseline and One month
  Vascular congestion will be evaluated using VExUS (Volume Evaluation by UltraSound)
Change in left ventricular filling pressures | Baseline and One month
  Left ventricular filling pressures to measure vascular and will be evaluated using the echocardiographic parameter E/e' (surrogate of LV filling pressures)
Change in plasma concentrations of catecholamines | Baseline and One month
  Neurohormonal activation to measure vascular congestion and will be evaluated using plasma concentrations of catecholamines.
Change in plasma concentrations of aldosterone | Baseline and One month
  Neurohormonal activation to measure vascular congestion and will be evaluated using plasma concentrations of aldosterone.
Change in plasma concentrations of plasma renin activity | Baseline and One month
  Neurohormonal activation to measure vascular congestion and will be evaluated using plasma concentrations of plasma renin activity

CONTACTS AND LOCATIONS:
Overall Officials: Carlos G Santos-Gallego, MD, Principal Investigator — Icanh School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 9 months and ending 36 months following article publication.